CLINICAL TRIAL: NCT04391699
Title: Humidifier Study: Evaluation of Prophylactic Heated Humidification on Obstructive Sleep Apnea (OSA) Patient Short Term Compliance to CPAP Therapy: Randomized Clinical Trial
Brief Title: Evaluation of Prophylactic Heated Humidification on Obstructive Sleep Apnea (OSA) Patient Short Term Compliance to CPAP Therapy
Acronym: Humidifier
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: cancelled before initiation
Sponsor: ResMed (Industry)
Collaborators: DOM AIR (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Humidifier 001
Record Dates: First submitted 2018-01-29; First posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Osa Syndrome
MeSH Terms: conditions — Carnevale syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP + Heated humidification (Experimental): CPAP + Heated humidification
  Interventions: Device: heated humidification
- CPAP alone (No Intervention): CPAP

INTERVENTIONS:
Device: heated humidification — heated humidification system
  Arms: CPAP + Heated humidification

SUMMARY:
To compare two different clinical strategies in order to evaluate the impact of prophylactic heated humidification on OSA patients' compliance to CPAP therapy.

DETAILED DESCRIPTION:
To compare two different clinical strategies in order to evaluate the impact of prophylactic heated humidification on OSA patients' compliance to CPAP therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patient
* Newly diagnosed OSA Patients eligible to CPAP therapy
* Signed informed consent

Exclusion Criteria:

* CPAP therapy contraindications
* Pregnancy
* Patient unable to come to study follow up visits or unable to finish the study.
* Informed consent not signed
* Adults who are subject to a legal protection measure or are unable to express their consent (such as patients under guardianship and patients deprived of judicial or administrative freedom)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
CPAP mean usage (hours/night) at the 3 month follow up | 3 months
  therapy compliance

SECONDARY OUTCOMES:
Sleep quality | 3 months
  pittsburgh sleep questionnaire index. total score
sleepiness | 3 months
  epworth sleep scale. total score

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Raymond, MD, Principal Investigator — clinique Bel Air
Locations (1):
- Clinique Bel Air, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No